CLINICAL TRIAL: NCT01324596
Title: A Randomised Evaluation of Molecular Guided Therapy for Diffuse Large B-cell Lymphoma With Bortezomib
Acronym: REMoDL-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHMCAN0749
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Lymphoma, Large B-Cell, Diffuse; Bortezomib; R-CHOP; Molecular profiling; Chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: R-CHOP (Active Comparator): Participants receive 6 cycles of conventional R-CHOP chemotherapy on a standard 21 day schedule: Rituximab 375mg/m2 intravenous Cyclophosphamide 750mg/m2 Intravenous Doxorubicin 50mg/m2 Intravenous Vincristine intravenous Prednisolone 100mg od orally
  Interventions: Drug: Intravenous
- Arm B: RB-CHOP (Experimental): Participants in this arm will receive 1 cycle of conventional R-CHOP chemotherapy, followed by 5 cycles of R-CHOP:
  Cyclophosphamide 750mg/m2 Intravenous Doxorubicin 50mg/m2 Intravenous Vincristine intravenous bortezomib - Intravenous Prednisolone 100mg od orally
  .
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Intravenous — Chemoimmunotheraphy
  Other Names: Rituximab; cyclophosphamide; doxorubicin; vincristine; prednisolone
  Arms: Arm A: R-CHOP
Drug: Bortezomib — Chemoimmunotheraphy
  Other Names: rituximab; cyclophosphamide; doxorubicin; vincristine; prednisolone
  Arms: Arm B: RB-CHOP

SUMMARY:
The aims of this study are:

* To evaluate the benefits of the addition of bortezomib to standard rituximab with cyclophosphamide, doxorubicin, vincristine, prednisolone (R-CHOP) therapy in Diffuse Large B-cell Lymphoma (DLBCL).
* To determine whether molecular phenotype effects the benefits derived from the addition of bortezomib.

DETAILED DESCRIPTION:
REMoDLB is a trial which aims to determine whether the addition of bortezomib (a drug that blocks the action of cellular complexes that break down proteins) to standard combination chemotherapy (called R-CHOP) improves how long patients with diffuse large B cell lymphoma survive without a recurrence of the disease. Results from recent research have suggested that patients can be divided into two biologically distinct subgroups labeled GCB (germinal centre derived B-cells like) and ABC (activated peripheral B-cells like).

GCB patients tend to do well with standard combination chemotherapy, but ABC patients have the majority of treatment failures. It is thought that ABC patients will benefit most from the addition of bortezomib.

The trial will be discussed with the patient. They will be asked to consent to molecular profiling of their tumour block whilst they have some time to consider whether they wish to enter the main trial. This will allow more time for this sample to be analysed and their particular biological subgroup to be determined.

All patients consenting to enter the main study will be given an initial cycle of RCHOP chemotherapy. Within each subgroup (ABC or GCB) patients will be randomly assigned to receive either RCHOP or RCHOP and bortezomib to ensure that the same number of each biological subgroup will receive the two treatments. All patients will then have 5 cycles of their assigned treatment regimen (either RCHOP or RCHOP and bortezomib). All patients will be followed up for a period of five years once they have completed their chemotherapy. The GCB group receiving RCHOP and bortezomib will be regularly checked to see if the new treatment is improving survival without recurrence of the disease. If the addition of bortezomib is not found to be beneficial for this group of patients this part of the trial will be stopped and all GCB patients will receive the standard treatment only (RCHOP).

It is anticipated that between 560 and 892 patients will be randomly allocated to the two treatments, the exact number depends on whether the GCB group receiving RCHOP and bortezomib is stopped or not.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL, expressing CD20. Sufficient diagnostic material should be available to forward to Haematological Malignancies Diagnostic Service (HMDS) for gene expression profiling and central pathology review. Core biopsies are acceptable, however the molecular profiling success rate is inferior compared to larger surgically acquired tissue samples. Best diagnostic practice encourages investigators to seek the latter approach whenever clinically appropriate.
* Measurable disease of at least 15mm.
* Not previously treated for lymphoma and fit enough to receive combination chemoimmunotherapy with curative intent.
* Age > 18 years.
* Stage IAX (bulk defined as lymph node diameter > 10cm) to stage IV disease and deemed to require a full course of chemotherapy.
* ECOG performance status 0-2.
* Adequate bone marrow function with platelets > 100x109/L; neutrophils >1.0x109/L at study entry, unless lower figures are attributable to lymphoma.
* Serum creatinine < 150μmol/L, measured or calculated creatinine clearance > 30mls/min, serum bilirubin < 35μmol/L and transaminases < 2.5x upper limit of normal at the time of study entry, unless attributable to lymphoma.
* Cardiac function sufficient to tolerate 300mg/m2 of doxorubicin. A pre-treatment echocardiogram is not mandated, but recommended in patients considered at higher risk of anthracycline cardiotoxicity.
* No concurrent uncontrolled medical condition.
* Life expectancy > 3 months.
* Adequate contraceptive precautions for all patients of child bearing potential.
* A negative serum pregnancy test for females of child bearing potential or those < 2 years after the onset of the menopause.
* Patients will have provided written informed consent.

Exclusion Criteria:

* Previous history of treated or untreated indolent lymphoma. However newly diagnosed patients with DLBCL who are found to also have small cell infiltration of the bone marrow or other diagnostic material (discordant lymphoma) will be eligible.
* Diagnosis of primary mediastinal lymphoma
* Uncontrolled systemic infection.
* History of cardiac failure of uncontrolled angina.
* Clinical CNS involvement.
* Serological positivity for Hepatitis C, B or known HIV infection. Viral serological testing is not mandated for study entry, but considered standard of care. (• Positive test results for chronic HBV infection (defined as positive HBsAg serology) will not be eligible. • Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) will not be eligible as one would normally monitor HBV DNA serially and add lamivudine if copy number became detectable. There is an interaction between lamivudine and bortezomib. Reactivation of latent infection has been reported with the use of bortezomib in this population (along obviously with the well recognised reactivation following R-CHOP). For these patient safety reasons, these patients should be excluded. • Patients who have protective titres of hepatitis B surface antibody (HBSAb) after vaccination are eligible. • Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing) will not be eligible.)
* Serious medical or psychiatric illness likely to affect participation or that may compromise the ability to give informed consent.
* Active malignancy other than fully excised squamous or basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix in the preceding 5 years.
* History of allergic reaction to substances containing boron or mannitol.
* Patient unwilling to abstain from green tea and preparations made from green tea as bortezomib may interact with these.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1132 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Event-free survival | 5 years
Disease-free survival | 5 years
Time to progression | 5 years
Response duration | 5 years
Complete and overall response rates | 5 years
Evaluation of toxicity (according to CTCAE version 4.0) | 5 years
Quality of life and assessment of peripheral neuropathy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Prof Peter Johnson, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (109):
- Switzerland (13):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Liestal, Basel
  - Universitatsspital Basel, Basel
  - Ospedale Regionale Bellinzona e Valli (IOSI), Bellinzona
  - Inselspital Bern, Bern
  - STSAG Thun, Bern
  - Spitalzenturm Oberwallis, Brig
  - Kantonsspital Graubunden, Chur
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich
  - UniversitatsSpital Zurich, Zurich
- United Kingdom (96):
  - University Hospital Aintree, Aintree
  - Monklands, Hairmyres and Whishaw Hospitals, Airdrie
  - Antrim Area Hospital, Antrim
  - Stoke Mandeville Hospital and Wycombe Hospital, Aylesbury
  - Ysbyty Gwynedd Hospital, Bangor
  - Basildon Hospital, Basildon
  - North Hampshire & Basingstoke Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Belfast City Hospital, Belfast
  - Arrowe Park, Birkenhead
  - Good Hope Hosptial, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Sandwell General Hospital Birmingham, Birmingham
  - Victoria Hospital, Blackpool
  - Royal Bournemouth, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Queen's Hospital Burton, Burton-on-Trent
  - West Suffolk Hospital, Bury St Edmunds
  - Velindre Hospital, Cardiff
  - Broomfield Hospital, Chelmsford
  - Cheltenham General Hospital and Gloucestershire Royal Infirmary, Cheltenham
  - Chesterfield Royal, Chesterfield
  - St Richard's Hospital, Chichester
  - Colchester General Hospital, Colchester
  - University Hospital Coventry, Coventry
  - Darent Valley Hospital, Dartford
  - Royal Derby Hospitals, Derby
  - Doncaster Royal Infirmary, Doncaster
  - Ulster Hospital, Dundonald
  - Royal Devon and Exeter Hospital, Exeter
  - Queen Elizabeth Hospital, Gateshead, Gateshead
  - Medway Maritime Hospital, Gillingham
  - Beatson West of Scotland Cancer centre, Glasgow
  - Diana Princess of Wales, Grimsby, Grimsby
  - Harrogate District Hospital, Harrogate
  - Hemel Hempstead General and Watford General, Hemel Hempstead and Watford
  - Huddersfield Royal Infirmary, Huddersfield
  - Castle Hill Hospital, Hull
  - Raigmore Hospital, Inverness
  - Kent and Canterbury Hospital, Kent
  - Queen Elizabeth Hospital, Kings Lynn
  - St James University Hospital, Leeds
  - Lincoln County Hospital, Pilgrim Hospital, Grantham and District Hospital, Lincoln
  - Royal Liverpool, Liverpool
  - Barnet General Hospital, London
  - Ealing Hospital, London
  - Guy's Hospital, London
  - Hammersmith Hospital, London
  - Hillingdon Hospital, London
  - King's College Hospital, London
  - Northwick Park Hospital, London
  - Princess Royal University Hospital, London
  - QE Woolwich, London
  - Royal Free Hospital, London
  - St Bartholomews Hospital, London
  - St George's Hospital, London
  - St Helier Hospital, London
  - The Royal Marsden, London
  - University College Hospital London, London
  - Luton and Dunstable Hospital, Luton
  - Maidstone Hospital and The Tunbridge Wells Hospital, Maidstone
  - Christie Hospital, Manchester
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Milton Keynes General Hospital, Milton Keynes
  - Freeman Hospital, Newcastle, Newcastle
  - Northampton General Hospital, Northampton
  - Mount Vernon Hospital, Northwood
  - Nottingham City Hospital, Nottingham
  - George Eliot Hospital, Nuneaton
  - Royal Oldham, Oldham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Poole General Hospital, Poole
  - Craigavon Area Hospital, Portadown
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire Hospital, Reading
  - Glan Clwyd District General Hospital, Rhyl
  - Queen's Hospital, Romford
  - Salisbury District Hospital, Salisbury
  - Scunthorpe General Hospital, Scunthorpe
  - Royal Hallamshire Hospital, Sheffield
  - Wexham Park, Slough
  - Southampton General Hospital, Southampton
  - Southend Hospital, Southend
  - County Hospital, Stafford
  - Royal Stoke Hospital, Stoke
  - Sunderland Royal Hospital, Sunderland
  - Great Western Hospital, Swindon
  - Torbay District General Hospital, Torbay
  - Royal Cornwall Hospital, Truro
  - Pinderfields Hospital, Dewsbury Hospital and Ponerfract Hospital, Wakefield
  - Warwick Hospital, Warwick
  - Worcestershire Royal Hospital, Worcester
  - Worthing Hospital, Worthing

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Davies AJ, Barrans S, Stanton L, Caddy J, Wilding S, Saunders G, Mamot C, Novak U, McMillan A, Fields P, Collins GP, Stephens R, Cucco F, Sha C, van Hoppe M, Tooze R, Davies JR, Griffiths G, Schuh A, Burton C, Westhead DR, Du MQ, Johnson PWM. Differential Efficacy From the Addition of Bortezomib to R-CHOP in Diffuse Large B-Cell Lymphoma According to the Molecular Subgroup in the REMoDL-B Study With a 5-Year Follow-Up. J Clin Oncol. 2023 May 20;41(15):2718-2723. doi: 10.1200/JCO.23.00033. Epub 2023 Mar 27. PMID 36972491
- [Derived] Davies A, Cummin TE, Barrans S, Maishman T, Mamot C, Novak U, Caddy J, Stanton L, Kazmi-Stokes S, McMillan A, Fields P, Pocock C, Collins GP, Stephens R, Cucco F, Clipson A, Sha C, Tooze R, Care MA, Griffiths G, Du MQ, Westhead DR, Burton C, Johnson PWM. Gene-expression profiling of bortezomib added to standard chemoimmunotherapy for diffuse large B-cell lymphoma (REMoDL-B): an open-label, randomised, phase 3 trial. Lancet Oncol. 2019 May;20(5):649-662. doi: 10.1016/S1470-2045(18)30935-5. Epub 2019 Apr 1. PMID 30948276